CLINICAL TRIAL: NCT07028255
Title: Effectiveness of Qualia Testosterone Supplementation on Testosterone Levels: A Randomized Double-Blind Parallel Trial
Brief Title: Effectiveness of Qualia Testosterone Supplementation on Testosterone Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qualia Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: QLS-013
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Testosterone
Keywords: testosterone supplementation; testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qualia Testosterone (Active Comparator): Qualia Testosterone manufactured by Qualia Life Sciences
  Interventions: Dietary Supplement: Qualia Testosterone
- Placebo (Placebo Comparator): Rice Flour
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Qualia Testosterone — Qualia Testosterone manufactured by Qualia Life Sciences
  Arms: Qualia Testosterone
Dietary Supplement: Placebo — Rice Flour
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled parallel trial designed to assess the efficacy of Qualia Testosterone, a novel dietary supplement, in adult males aged 28 to 65 experiencing symptoms associated with testosterone deficiency. Approximately 60 participants will be randomized to receive either Qualia Testosterone (2 capsules daily) or a matched placebo for 21 days, with dosing administered each morning. The study's primary outcomes are changes in total testosterone, free testosterone (via dialysis), and dihydrotestosterone levels from baseline to Week 3. Secondary outcomes include changes in Aging Male Symptoms Scale scores-encompassing psychological, somatic, and sexual domains-as well as safety and tolerability. Blood samples will be collected in a laboratory setting, while symptom and safety assessments will be completed electronically at home.

ELIGIBILITY:
Inclusion criteria:

Provide voluntary, written, informed consent to participate in the study Agree to provide a valid cell phone number and are willing to receive communications through text Can read and write English Willing to not begin taking any new supplements during the study and continue taking any supplements they are currently using regularly Willing to complete questionnaires, records, and diaries associated with the study.

Male participants aged 28-65 A score ≥27 on the Aging Males Symptom Scale Willing and able to visit a local blood draw facility for required blood sample collections Live within 20 miles of a suitable blood draw facility Willing to not consume any supplements containing Testosterone starting about 2 weeks prior to the baseline blood test test continuing through the intervention period.

Exclusion criteria:

Known food intolerances/allergy to any ingredients in the product Having any of the following conditions: Psychiatric conditions, neurologic disorders, endocrine disorders, cancer Having had a significant cardiovascular event in the past 6 months Taking MAO inhibitors, SSRIs, or any other psychiatric or neurological medicines On immunosuppressive therapy Individuals who were deemed incompatible with the test protocol Adults lacking capacity to consent Have Hypogonadism

Ages: 28 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Between-group change in blood testosterone levels | 3 weeks
  To assess the between-group differences in change from baseline to Week 3 in Total Testosterone, Free (Dialysis) Testosterone, and Dihydrotestosterone levels following Qualia Testosterone supplementation.

SECONDARY OUTCOMES:
Aging Male Symptoms Scale scores | Week 3
  To evaluate between-group changes in Overall, Psychological, Somatic, and Sexual scores on the Aging Male Symptoms Scale from baseline to Week 3
Side effect profile as measured by a custom Safety and Tolerability survey | Week 1, 2 and 3
  Number of participants with treatment-related adverse events as assessed by a score of 3 or greater on the Safety and Tolerability survey

CONTACTS AND LOCATIONS:
Locations (1):
- Qualia Life Sciences, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No